CLINICAL TRIAL: NCT07203209
Title: No Additional Benefits of Thoracic Mobility Exercises in Addition to Training on Different Athletic Skills of Adolescent Volleyball Players: A Randomized Controlled Study
Brief Title: Thoracic Mobility Exercises on Athletic Skills of Adolescent Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, özge ece günaydın, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-FTR-EG-03
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Thoracal Mobility
Keywords: exercise; thoracal mobility; volleyball player; adolescents
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracal mobility group (Experimental): The participants allocated to this group will perform thoracal mobility exercises added to regular training for 4 weeks.
  Interventions: Other: thoracal mobility exercises
- Control group (Other): The participants allocated to this group will perform regular training program for 4 weeks.
  Interventions: Other: regular training

INTERVENTIONS:
Other: thoracal mobility exercises — The exercise program given to the athletes in the mobility group will include 8 exercises specially designed for thoracic region mobility. The exercises will be practiced by the team trainer in every training session and otherwise at home twice a day.
  Arms: Thoracal mobility group
Other: regular training — This training program is composed of the teams daily practice exercises.
  Arms: Control group

SUMMARY:
Thoracic mobility is a significant contributing factor to the enhancement of athletic abilities and performance. The aim of this study was to determine the effects of thoracic mobility exercises on strength, endurance, flexibility, and spike and serve speed of female adolescent volleyball players. Thirty-six adolescent female volleyball players will participate and be divided into two groups: one will receive regular training, while the other will receive additional thoracic mobility exercises for four weeks. Shoulder's Internal and external rotation strength, endurance, thoracic mobility, and spike and serve speeds will be evaluated.

DETAILED DESCRIPTION:
The ability of the shoulder and upper extremity to move in a functional manner is dependent upon the coordinated action of multiple body parts, including the shoulder, thoracic spine, and pelvis, which collectively form the kinetic chain. The kinematic relationship of the thoracic spine and shoulder within this synergy has not been fully explained. An understanding of kinematics allows for a comprehensive evaluation of the trunk position, which is a combination of thoracic and lumbar motion. This evaluation must consider the thoracic spine, as it also affects shoulder muscle function. Thoracic spine movement contributes to upper extremity functionality, especially in activities involving positions from the middle to the end of the shoulder range of motion in the sagittal plane. Therefore, deficiencies in thoracic extension may create more stress on other components of the kinetic chain in athletes engaged in overhead sports activities and may have a negative effect on the athlete's performance and ability to compete. Although the thoracic spine has not been covered much in the sports literature due to relatively low pain prevalence and measurement difficulties, evidence supports that the thoracic spine plays an important role in sports performance. An estimated 55% of the total force and kinetic energy generated during a throwing motion is of kinematic importance for the upper extremity, as it contributes approximately 80% of the total available trunk rotation motion. The incidence of elbow and shoulder injuries is three times higher in athletes with a limited range of motion in trunk rotation. Current rehabilitation approaches following shoulder injuries focus on treating the specific signs and symptoms of shoulder pathology rather than the possible disorders within the kinetic chain and the functional interaction between the shoulder complex and the trunk. Nevertheless, the incorporation of injury prevention and therapeutic modalities comprising thoracic mobility exercises into rehabilitation protocols is purported to be advantageous in terms of both athletic performance and the risk of recurrent injury to the elbow and shoulder regions.It is important to add thoracic mobility exercises to training at an earlier period to reduce upper extremity injury rates in elite athlete populations and to gain the practice habits of preventive exercises. If the spine, which is still undergoing development in adolescent athletes, can be trained in the direction of these gains, it is possible to achieve healthier athletes with a low incidence of injury and high levels of sporting performance. In the light of this literature information, the aim of this study was to investigate the effects of thoracic mobility exercises added to the training programs of adolescent volleyball players on shoulder strength, endurance, thoracic joint mobility and performance indicators such as spike and serve speeds. This study is designed as a randomized controlled study. For the athletes invited to the study, first randomization will be applied with computer-based program, and two groups will be formed as mobility and control. Then, thoracic rotation range of motion, trunk hyperextension levels, internal and external rotation muscle strengths, scapular endurance, spike and serve speeds and demographic data of all participants will be recorded. The control group participated only in team training while the mobility group will be subjected to thoracic mobility exercises in addition to team training for 4 weeks. The measurements will be repeated after 4 weeks to evaluate possible differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* being a female volleyball player between the ages of 13-17,
* being currently in a team
* participating in volleyball training for 2 hours at least 3 days a week.

Exclusion Criteria:

* musculoskeletal injuries of the neck, upper and lower extremities,
* orthopedic diseases
* being received physical therapy involving the shoulder and neck region in the last 6 months

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Due to hormonal changes during puberty, the musculoskeletal characteristics of boys and girls can differ. Therefore, we want our groups to be homogeneous, so we included girls' volleyball players.
Enrollment: 26 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Spike and serve speed | At the begining of the study and at th 4th week
  The serve and spike speeds of the volleyball players participating in the study will be evaluated with Pocket radar system.The highest serve and spike speeds will be included in the evaluation.
thoracolumbar rotation angle | at the begining of the study and at the 4th week
  Thoracolumbar rotation angle will be evaluated using a goniometer. Prior to the examination, the participants will be instructed for the correct movement technique in order to prevent the occurrence of compensatory movements in the shoulder and trunk.The athlete will perform trunk rotation first to the left and then to the right. At the last point, the rotation angle will be measured.

SECONDARY OUTCOMES:
Scapular muscle endurance | At the begining of the study and at the 4th week.
  Shoulder muscle endurance will be evaluated with the scapular muscle endurance test. The test will be performed with the players standing, facing the wall with their shoulders and elbows in the 90° flexion position.
shoulder strength | At the begining of the study and at the 4th week.
  The strength of the shoulder external and internal rotation muscles of the athlete will be evaluated using a digital hand dynamometer (Lafayette Instrument Company, USA) in a seated position on a chair with back support.
Trunk hyperextention | At the begining of the study and at the 4th week.
  Trunk hyperextension measurements of the subjects will be made with a tape measure. The athlete will be asked to touch the wall with his/her trunk by opening both feet in full external rotation with his/her face to the wall. In this position, the initial measurement will be taken between the sternum and the wall.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No